CLINICAL TRIAL: NCT05704153
Title: Modelling and Control of Non-invasive Vagus Nerve Stimulation for Autoimmune Diseases (1A)
Acronym: VaNeSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Universitat de Girona (Other); Hospital Mutua de Terrassa (Other); Imperial College London (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Judith Navarro, MD PhD, Consultant Neurologist, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: PID2020-117171RA-I00-1A
Record Dates: First submitted 2022-10-04; First posted 2023-01-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Systemic Lupus Erythematosus; Autoimmune Disorder; Vagus Nerve Autonomic Disorder
Keywords: Parasympathetic Nervous System; Vagus Nerve Stimulation
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: VaNeSA is a multicentre, national, randomized, double-blind, parallel-group, placebo-controlled, outpatient study.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Sham (Sham Comparator): Control group to be subjected to sham stimulation.
  Interventions: Device: Sham Intervention
- 30 hertz (Hz) Stimulation (Experimental): Group of patients treated via 30Hz transcutaneous electrical nerve stimulation
  Interventions: Device: Parasym 30Hz
- 1Hz Stimulation (Experimental): Group of patients treated via 1Hz transcutaneous electrical nerve stimulation
  Interventions: Device: Parasym 1Hz

INTERVENTIONS:
Device: Parasym 1Hz — Transcutaneous auricular vagus nerve stimulation of 1Hz
  Arms: 1Hz Stimulation
Device: Parasym 30Hz — Transcutaneous Auricular Vagus Nerve Stimulation of 30Hz
  Arms: 30 hertz (Hz) Stimulation
Device: Sham Intervention — Sham stimulation
  Arms: Sham

SUMMARY:
The overall goal of this clinical trial is to evaluate the causality relationship between the non vagus nerve stimulation waveform parameters and the therapeutic effect. Thus, unlocking a pathway to optimize parameters that maximize the benefits of therapy and minimize unwanted side effects. The experimental design includes the analysis of physiological signals, clinical biomarkers of disease, and clinical outcomes to determine the most effective measures for the monitoring, optimization, and personalization of non vagus nerve stimulation in systemic lupus erythematosus disease.

ELIGIBILITY:
Inclusion Criteria:

* Systemic lupus erythematosus (SLE) (defined by the American College of Rheumatology- or SLICC criteria)
* Musculoskeletal pain ≥ 4 on a non-anchored VAS 10 cm scale
* BILAG C on Musculoskeletal Domain of the BILAG 2004
* If on corticosteroids, the dose must be stable and ≤ 10mg/day (prednisone or equivalent) for at least 28 days before baseline,
* If on background immunosuppressive treatment the dose must be stable for at least 28 days before baseline
* Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

* Treatment with rituximab within one year of baseline as it is related to lymphocyte depletion that could alter the result of the biomarker study (subjects with previous treatment with rituximab can enter study only with documentation of B cell repletion).
* Treatment with cyclophosphamide within 2 months of baseline as it is related to lymphocyte depletion that could alter the result of the biomarker study.
* Expectation to increase steroids and/or immunosuppressive treatment.
* Anti-phospholipid syndrome.
* Fibromyalgia (fibromyalgia will be defined as a score > 13 on the Fibromyalgia Symptom Scale), chronic fatigue syndrome.
* Treatment with an anti-cholinergic or sympathicomimetic medication, including over the counter medications.
* Implantable electronic devices such as pacemakers, defibrillators, hearing aids, cochlear implants or deep brain stimulators.
* Joint replacement within 60 days prior to study enrolment or planned within the course of the study.
* Any planned surgical procedure requiring general anaesthesia within the course of the study.
* Intra-articular cortisone injections within 28 days of the start of study.
* Chronic inflammatory disorders apart from SLE affecting the joints.
* Investigational drug and/or treatment during the 28 days or seven half-lives of the investigational drug prior to the start of study drug dosing (Day 0), whichever is the greater length of time.
* Active infection including hepatitis B, hepatitis C or HIV at baseline due to high prevalence of neuropathy.
* Any condition which, in the opinion of the investigator, would jeopardize the subject's safety following exposure to a study intervention.
* Pregnancy or lactation.
* Haemoglobin below 9.0 gm/dL (by the most recent CBC) as anaemia is related to no- neurogenic orthostatic hypotension and increases cardiovascular symptoms in COMPASS 31 scale
* Comorbid disease that may require administration of corticosteroid use.
* Inability to comply with study and follow-up procedures.
* Known cardiac arrhythmia, severe cardiac disease or neurodegenerative disease.
* Known or confirmed at baseline screening peripheral or autonomic nervous system involvement, including LES-related, toxic polyneuropathies, metabolic neuropathies (including diabetes), etc.
* Previous experience with vagus nerve stimulation devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Systemic Lupus Erythematosus with clinical and analytic change after non-invasive vagus nerve stimulation (nVNS) at different waveform parameters | Visit 1(baseline, exploratory study, up to 30days prior to first nVNS)
  We will develop an nVNS platform with an integrated nVNS decision support system, including nVNS and physiological wearable sensors, that will optimize nVNS waveform parameters to maximize the therapeutic effect while minimizing unwanted side effects. Therapeutic effect and side effects will be measured by clinical, neurophysiological and analytic tests as described in "secondary outcome measures".

SECONDARY OUTCOMES:
Blood count | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Complete blood count
Erythrocyte sedimentation rate | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Marker of inflammatory conditions, mm/h
C-reactive protein | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Markers of inflammatory conditions, mg/dl
Anti-dsDNA | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Serological marker of activity in Systemic lupus erythematosus (SLE) ui/ml
C3, C4 | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Serological markers of activity in Systemic lupus erythematosus (SLE) g/l
Tumoral necrosis factor (TNF), Interleukin (IL) -6, IL-10 and Il1B | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Levels of pro-inflammatory cytokines, pg/ml
High mobility group box 1 protein (HMGB1) | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Levels of pro-inflammatory cytokines, ui
Alpha interferon (IFNα) | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Ratios of IFNα protein, ui
EuroQol-5D (EQ-5D-5L), | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels and 1 month after nVNS.
  EQ-5D-5L questionaries. Minimum 1, maximum 3, higher scores mean a worse outcome.
Lupus Patient-Reported Outcome (LupusPRO) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Lupus PRO questionaries. Minimum 0, maximum 5, higher scores mean a worse outcome.
Lupus Quality of Life (LupusQoL) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Lupus QoL questionaries. Minimum 1, maximum 7, higher scores mean a worse outcome.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  FACIT-F scale. Minimum 0, maximum 4, higher scores mean a worse outcome.
Fatigue Severity Scale (FSS) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  FSS. Minimum 1, maximum 7, higher scores mean a worse outcome.
Composite Autonomic Symptom Score (Compass-31) | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Self-scoring Compass 31 autonomic assessment. Minimum 0, maximum 100, higher scores mean a worse outcome.
28-joint count | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  28-joint count will be used to assess articular involvement.
Physician's Global Assessment (PGA) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  PGA as non-specific activity scale. Minimum 0, maximum 3, higher scores mean a worse outcome.
Patients' Global Assessment (PtGA) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  PtGA as non-specific activity scale. Minimum 0, maximum 100, higher scores mean a worse outcome.
Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  CLASI will be used to evaluate skin involvement.Minimum 0, maximum 100, higher scores mean a worse outcome.
Numeric scale ranges (NRS) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  11-point NRS scale for pain. Minimum 0, maximum 10, higher scores mean a worse outcome.
Visual Analog Scale (VAS) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  VSA for pain. Minimum 0, maximum 10, higher scores mean a worse outcome.
High-frequency power, low-frequency power | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Continuous electrocardiogram will be recorded at rest for 5 minutes for heart rate variability (HRV) analysis (high-frequency power HF, low-frequency power LF), m2
LF to HF power ratio | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Continuous electrocardiogram will be recorded at rest for 5 minutes for heart rate variability (HRV) analysis ( LF to HF power ratio)
Cardiovagal evaluation. (Composite autonomic scoring scale) | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Continuous electrocardiogram heart rate changes during deep breathing and postural changes (beats per minute).Composite autonomic scoring scale minimun 0, maximum 3, higher scores mean a worse outcome.
Vasalva ratio | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Continuous electrocardiogram heart rate changes during Valsalva manoeuvre (ratio).
Sympathetic evaluation (Composite autonomic scoring scale) | Baseline, after five days of stimulation and 1 month after stimulation. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Beat-to-beat blood pressure changes to isometric exercise, Valsalva manoeuvre and postural changes, (mmHg). Composite autonomic scoring scale minimun 0, maximum 4, higher scores mean a worse outcome.
Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Disease-specific activity scale. Minimum 0, maximum 105, higher scores mean a worse outcome.
BILAG-2004 | Baseline, days 1-2-3-4-5 of nVNS, after five days of nVNS, after 2 weeks of nVNS, after3 weeks of nVSN. Additionally, 2 and 3months after stimulation if the biomarkers and scales of activity do not return to baseline levels
  Disease-specific activity scale. Minimum 0, maximum 32, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Contreras I, Navarro-Otano J, Rodriguez-Pinto I, Guemes A, Alves E, Rios-Garces R, Espinosa G, Alejaldre A, Beneyto A, Ramkissoon CM, Vehi J, Cervera R. Optimizing Noninvasive Vagus Nerve Stimulation for Systemic Lupus Erythematosus: Protocol for a Multicenter Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 13;12:e48387. doi: 10.2196/48387. PMID 37831494
- See also: Framework of the general project lead by Iván Contreras : VaNeSA — https://micelab.udg.edu/projects/